CLINICAL TRIAL: NCT02884310
Title: Interest of the Gradient of Nociceptive Indexes After a Tetanus (100 Hz, 60 Milliamperes, 30 Seconds) at a Fixed Remifentanil Effect Site Concentration to Adjust Remifentanil Before Tracheal Intubation and Skin Incision
Brief Title: Interest of a Tetanus Test at a Fixed Remifentanil Concentration Before Laryngoscopy and Skin Incision
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Collaborators: University of Liege (Other)
Responsible Party: Principal Investigator, Luc Barvais, Professor and head of the cardiothoracic and vascular anesthesia Clinics, Erasme University Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: ErasmeUH P2012/20
Record Dates: First submitted 2016-08-18; First posted 2016-08-31 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Intravenous Anesthetic Agent Overdose
Keywords: Remifentanil; Heart Rate Variability; Pupil dilation; SPI
MeSH Terms: conditions — Mydriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SPI group (Experimental): Remifentanil titration before tracheal intubation and skin incision according to the SPI gradient obtained after a nociceptive test using a tetanic stimulus of 100 Hz, 60 milliamperes during 30 seconds performed at a 3 ng/ml level of the remifentanil concentration.
  During surgery, the effect site remifentanil concentration was either increased or decreased by 1 ng/ml to maintain SPI below 40 or above 20, respectively.
  Interventions: Drug: Remifentanil adapted to SPI
- Control group (Active Comparator): The remifentanil concentration before tracheal intubation and skin incision was fixed at 4 ng/ml.
  During surgery, the remifentanil concentration was adapted according to the hemodynamic answer of the patient. It was changed by 1 ng/ml stepwise variations to maintain heart rate and mean blood pressure within 20% of the patient reference hemodynamic values.
  Interventions: Drug: Remifentanil fixed

INTERVENTIONS:
Drug: Remifentanil adapted to SPI
  Arms: SPI group
Drug: Remifentanil fixed
  Arms: Control group

SUMMARY:
Individually-tailored administration of the opioid analgesic component during general anaesthesia is still a challenge for the anesthesiologist. The aim of this protocol is to look if the gradient response of a nociception index to a calibrated tetanic stimulus during standard anesthetic conditions, could help to titrate remifentanil analgesia before tracheal intubation and before skin incision. The studied parameters are the SPI index developed by General Electric, the "Analgesia Nociception Index" and the pupil dilation using the pupil scan algometer.

DETAILED DESCRIPTION:
Two randomized groups of patients scheduled for general surgery under Target Controlled remifentanil propofol anaesthesia are compared.

All patients receive two standard calibration tests (Tetanic stimulus at the ulnar nerve: 100 Hertz, 60 milliamperes, 30 seconds) before tracheal intubation and skin incision at a stable remifentanil level of 3 ng/ml. Propofol concentration is targeted to maintain the BIS value as close as possible to 50. Patients are mechanically ventilated at an inspired O2 concentration of 50% and using tidal volumes of 8 to 10 mL/kg and respiratory rates of 12 to 15/min. Patients receive an induction dose of neuromuscular blocking agent.

In the treated group, the importance of the Surgical Plethysmogram Index (SPI) gradient after the tetanic stimulus will guide the subsequent administration of remifentanil to cover tracheal intubation and surgical incision. As compared to SPI value before the calibration test, a less than 10 unit increase in SPI will not prompt any change in remifentanil concentration before tracheal intubation and surgical incision. An increase in SPI between 10 and 20 units will prompt a remifentanil effect-site target concentration of 4 ng/ml, between 20 and 30 of 5 ng/ml, and above 30 of 6 ng/ml for tracheal intubation. Once the trachea is intubated, remifentanil concentration will be lowered to 3 ng /ml. It will be adjusted again before surgical incision according to the same criteria. Ten minutes after surgical incision until the end of the surgical procedure, the remifentanil concentration will be targeted to maintain SPI between 20 and 50.

In the control group, conditions will be the same as those of first group, except that remifentanil concentration will be adjusted according to heart rate and blood pressure. The anesthesiologist in charge is blinded to the results of the SPI gradient after the two calibration tests at 3 ng/ml remifentanil concentration and also blinded to the 2 other nociception indexes at all times. Remifentanil concentration is targeted at 4 ng/ml before tracheal intubation and surgical incision. Ten minutes after skin incision until the end of surgery, remifentanil concentrations will be adjusted according to the hemodynamic parameters.

Data acquisition and analysis will lead to the following statistical comparisons between the two groups:

* Hemodynamic reactivity to tracheal intubation and surgical incision.
* Concordance between SPI, Analgesia Nociception Index (ANI), and pupil diameter variations in response to the calibration test and during maintenance of anesthesia.
* Reliability of the prediction of hemodynamic reactivity to intubation and incision by the SPI, ANI, pupil diameter and hemodynamic response to the calibration test, and improvement of the prediction when combining the information given by those parameters.

2.2. Monitoring The monitoring will correspond to the classical monitoring of any general anesthesia procedures (Electrocardiogram, peripheral saturation in O2, Non-Invasive Blood Pressure, respiratory gases, pressure and flows in the airway, muscle relaxation).

The following parameters will be continuously recorded and saved for subsequent analysis :

* Heart rate
* Inspired and expired gases : O2, Carbon dioxide (CO2)
* Spirometry : peak, plateau, and end-expiratory pressures
* EKG : heart rate
* Non-invasive blood pressure : automatic measured every 5 minutes
* SPI

Additional monitoring :

* Bispectral Index (BIS)
* ANI
* Pupil dilation measurement

2.3. Anesthetic medications

2.3.1. Premedication The premedication will consist of 0.5 mg oral alprazolam (XANAX) one hour before induction of anesthesia.

2.3.2. Anesthesia General anesthesia will be induced and maintained using Target Controlled Infusions (TCI) of propofol and remifentanil, and using a single cisatracurium bolus.

2.3.2.1. Induction of anesthesia In the experimental group, the initial target effect-site concentration (Ce) of remifentanil will be 3 ng/ml and 3 µg/ml for propofol. The propofol Ce will be increased by steps of 1 µg/ml until loss of consciousness (6.0 µg/ml maximum). A 0.2 mg/kg bolus of cisatracurium will be given immediately after loss of consciousness. The tetanic calibration test will be performed once all responses to train of four (TOF) stimulation have disappeared. The BIS target before the tetanic stimulation will be 50 (range 40-60).

Pupil dilation and the ANI response to the tetanic stimulation will also be measured.

After tracheal intubation, remifentanil concentration will be reduced to 3 ng/ml, and propofol concentration adjusted to keep the BIS value as close to 50 as possible.

In the control group, the induction of anesthesia will occur the same way as in the experimental group, except that the initial concentration of remifentanil will be 3 ng/ml, and 4 ng/ml for tracheal intubation and incision. It will be changed according to hemodynamic parameters thereafter. Propofol concentration will be targeted to maintain stable BIS values around 50. The tetanic calibration test will be performed blindly once all responses to TOF stimulation have disappeared, and once propofol and remifentanil concentrations have been stable for more than 5 minutes. SPI, ANI, and pupil diameter values will be blindly recorded.

2.3.2.2. Maintenance of anesthesia The upper and lower limits of propofol concentrations will be 2.0 and 6.0 µg/ml, respectively. It will be targeted to maintain a stable BIS value around 50. During surgery, remifentanil concentrations will range between 2.0 and 10 ng/ml. In the experimental group (SPI), the calibration test-defined remifentanil concentration and the pre-incision propofol concentration will be kept intact for 10 minutes after the surgical incision. Thereafter, they will be modified according to the below-defined criteria.

In the control group, remifentanil concentration will be maintained at 4 ng/ml during 10 minutes after the surgical incision. Thereafter, propofol and remifentanil concentrations will be modified according to hemodynamic reactivity, and according to BIS, which will be kept at 50 (see tables below). SPI, and the other nociception indexes will be blindly recorded in that group.

2.3.2.3. Propofol concentration adaptations in both groups Propofol concentrations will be adapted to maintain BIS as close to 50 as possible. Changes in propofol concentration will be allowed every 5 minutes after having reached the new target, if necessary, as a function of criteria defined in Table 2.

Table 2 Propofol concentration adaptation as a function of BIS BIS Change in propofol concentration >70 +2 µg/ml > 55 +1 µg/ml < 45 -0.5 µg/ml < 35 -1 µg/ml

2.3.2.4. Remifentanil concentration adaptations

2.3.2.4.1. In the experimental group The goal in the experimental group will be to maintain a SPI value between 20 and 40 during surgery, from 10 minutes after incision to the end.

After incision, remifentanil concentration will be adapted according to criteria defined in Table 3.

Table 3 Remifentanil concentration adaptation during surgery (range 2 to 10 ng/ml) Event Change in remifentanil concentration SPI<20 -1 ng/ml SPI>50 +1 ng/ml SPI>80 +2 ng/ml

In case of hemodynamic reactivity (increase or decrease of more than 20 % as compared to reference values), despite adequate adaptation of remifentanil concentration as a function of SPI, it will be corrected according to criteria defined in paragraph 2.5 for hypotension or bradycardia episodes. In case of hypertension, (more than 20% as compared to reference value), despite adequate remifentanil concentration adaptation as a function of SPI, 0.5 mg intravenous boluses of nicardipine (Nicardipine) will be administered intravenously until return to acceptable values. Similarly, in case of tachycardia despite adequate adaptation of remifentanil adaptation as a function of SPI values, it will be corrected by 1 mg intravenous boluses of metoprolol (Seloken) until return to pre-defined values. In the event of both cases, exclusion of the patient's data from statistical analysis should be considered.

2.3.2.4.2. In the control group Before surgical incision, in the absence of hemodynamic reactivity, remifentanil concentration will be 4 ng/ml, and will not change for 10 minutes after incision.

Ten minutes after incision, remifentanil concentration will be adapted according to hemodynamic reactivity

Table 4 Remifentanil concentration adaptation in the Control group Hemodynamic Reactivity (> 20% as compared to reference values or Mean Arterial Pressure (MAP) > 90 mmHg and/or Heart Rate (HR) > 100/min): -1 ng/ml Hypotension/bradycardia (<20% as compared to reference values or MAP < 60 mmHg and/or HR < 45/min): +1 ng/ml

Remifentanil concentration will always be kept between 2 and 10 ng/ml. In case of hemodynamic changes at those concentrations, they will be corrected according to the criteria defined above for the SPI group.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Informed consent obtained during the pre-anesthetic visit
* American Society Anesthesiology status I or II
* Scheduled surgery under general anesthesia, and necessitating endotracheal intubation and controlled mechanical ventilation
* Body mass index (BMI) between 17 and 30 kg/m2

Exclusion Criteria:

* Pregnancy
* Patient refusal
* Pace maker (all modes)
* Heart failure

  * Ejection fraction < 50%
  * Symptomatic aortic or mitral pathology
* Non sinus rhythm
* Chronic use of beta blocking agents or other anti-hypertensive medications, except for diuretics
* Dysautonomia
* Diabetes
* Spontaneous ventilation during anesthesia
* Allergy to one of the medications used during this experiment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
hemodynamic stability following tracheal intubation and surgical incision | within 60 minutes after anesthesia induction
  Improvement of hemodynamic stability at anesthesia induction if remifentanil analgesia is not fixed at a predefined value for all patients but adapted to a nociceptive test at a predefined remifentanil concentration

SECONDARY OUTCOMES:
hemodynamic stability during surgery | within surgery
  Improvement of hemodynamic stability during surgery if remifentanil is adapted to SPI changes

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Defresne A, Barvais L, Clement F, Bonhomme V. Standardised noxious stimulation-guided individual adjustment of remifentanil target-controlled infusion to prevent haemodynamic responses to laryngoscopy and surgical incision: A randomised controlled trial. Eur J Anaesthesiol. 2018 Mar;35(3):173-183. doi: 10.1097/EJA.0000000000000742. PMID 29189318